CLINICAL TRIAL: NCT06829693
Title: Evaluation of the Incidence of Psychiatric Disorders As a Function of First-line Antiepileptic Drug Prescribing Practices: Use of Assurance Maladie Databases
Acronym: PRADOV
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government); GHU Paris Psychiatry & Neurosciences (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240983; PREPS 2024 - 983 (Other Grant/Funding Number: Ministry of health, France)
Record Dates: First submitted 2025-01-24; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Epilepsy; Side Effects of Drugs
Keywords: epilepsie; snds; bases de données médico-administratives
MeSH Terms: conditions — Epilepsy; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An estimated 600,000 people suffer from epilepsy in France, with a prevalence of around 0.6%. The disease and its associated co-morbidities, particularly psychiatric, have a detrimental effect on the patient's quality of life. Recommendations for the management of epilepsy are based primarily on antiepileptic drug treatment. Therapeutic recommendations for this management have a limited level of evidence (usually grade C or expert agreement), with very few high-level evidence recommendations (grade A or B). In the first instance, monotherapy with progressive doses is recommended to avoid adverse effects at the start of treatment, notably sedation and dizziness.

Levetiracetam is one of the most widely prescribed antiepileptic drugs, thanks to its broad spectrum of antiepileptic activity and its reputedly favorable safety profile. In practice, however, this drug is associated with sometimes severe psychobehavioral side effects, including irritability and insomnia, as well as psychiatric side effects such as manic episodes, depressive episodes and suicidal crises. These psycho-behavioral and psychiatric episodes are described in the literature in cohorts of patients monitored in expert centers. In contrast, there are few published data on a population scale in primary care. Moreover, the risk factors for psychobehavioral and psychiatric episodes on levotetracetam are insufficiently known, and there are few data in terms of impact on the safety of the care pathway. In addition to the development of psychiatric comorbidities, potential negative impacts on the patient's care pathway include interruptions in anti-epileptic treatment with the risk of therapeutic failure, increased healthcare consumption and, ultimately, a deterioration in the patient's quality of life.

As these psychiatric side-effects are not well known to the majority of general practitioners, who are the main primary prescribers of antiepileptic drugs, we can hypothesize that there are many patients for whom these psychiatric disorders are not attributed to the antiepileptic treatment, and that the latter is not modified, negatively impacting the safety of the care pathway. It is for this reason that the latest HAS report of March 23, 2023 recommends that the initiation of the first treatment be carried out on the recommendation of a neurologist. The main objective is to estimate, among patients with no psychiatric history, the risk of developing psychiatric disorders in the year following initiation of 1st-line antiepileptic treatment, as a function of (i) the treatment prescribed in 1st line and (ii) the sequence of treatments, i.e. the sequence of different antiepileptic treatments. It is a retrospective cohort on medico-administrative databases. The inclusion period is January 1, 2016 - December 31, 2023 and all adult patients (age ≥ 18 years), affiliated to the social security system with a first reimbursement of antiepileptic treatment is included.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (age ≥ 18 years), affiliated to the social security system with a first reimbursement of antiepileptic treatment

Exclusion Criteria:

* Patients with a psychiatric comorbidity, treated or not in the year preceding the index date of first prescription of the antiepileptic drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients benefiting from reimbursement by French health insurance for long-term antiepileptic treatment, and appearing in the health insurance reimbursement database.
Sampling Method: Non-Probability Sample
Enrollment: 355000 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
risk of developing psychiatric disorders in the year following initiation of 1st-line antiepileptic treatment | 12 months
  Incidence of psychiatric disorders 1 year after initiation of antiepileptic treatment, defined as :
  * Any hospitalization in MCO or RIM-P for psychiatric causes: ICD-10 codes F00 to F99 in DP or DR, except codes F70 to F79 (mental retardation) and F90 to F98 (behavioral and emotional disorders appearing during childhood and adolescence),
  * Any consultation with a city psychiatrist or hospital psychiatrist (as part of an outpatient procedure),
  * Any first prescription of a psychotropic drug: anxiolytics (ATC N05B*) - hypnotics (ATC N05C*) - antidepressants (ATC N06A*) - antipsychotics (ATC N05A*).

CONTACTS AND LOCATIONS:
Locations (1):
- European Georges Pompidou Hospital, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No
French law does not allow the sharing of data from the French insurance database.